CLINICAL TRIAL: NCT03084133
Title: Impact of EDUcation Strategy on Patients With COLorectal CANCER or Advanced Adenoma in the Detection of Colorectal Cancer of Their First-degree Relatives - Randomized, Multicenter Cluster Test
Brief Title: Impact of EDUcation Strategy on Patients With COLorectal CANCER or Advanced Adenoma in the Detection of Colorectal Cancer of Their First-degree Relatives
Acronym: EDUCANCOLAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Collaborators: University Hospital, Angers (Other Government); Nantes University Hospital (Other); Centre Hospitalier de Dreux (Other); Hospital BLOIS (Unknown); Hospital LOCHES (Unknown); Poitiers University Hospital (Other); UNIVERSITY HOSPITAL, ORLEANS (Unknown); Clinic LE MANS (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INCA14-TL/EDUCANCOLAGE; 2015-A01514-45 (Other: ID RCB)
Record Dates: First submitted 2017-02-28; First posted 2017-03-20 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Cancer Colorectal
Keywords: Therapeutic education strategy
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Intervention Model Description: "Intervention group" means a screening information and education system in which the particularities of the index cases likely to require adaptation of the device will be collected, analyzed and taken into account.
  "Control group": provision of information on the need for screening colonoscopy in first-degree relatives of case-index patients by the practitioner taking charge of the case-index according to its usual practice and adapted to the level of understanding of Case-index.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic Education Strategy (Experimental): Means a screening information and education system in which the particularities of the index cases likely to require adaptation of the device will be collected, analyzed and taken into account.
  Intervention 'Therapeutic Education Strategy'
  Interventions: Behavioral: Therapeutic Education Strategy
- Control group (No Intervention): Provision of information on the need for screening colonoscopy in first-degree relatives of case-index patients by the practitioner taking charge of the index case according to its usual practice

INTERVENTIONS:
Behavioral: Therapeutic Education Strategy — In the experimental arm of the study ("intervention group"), a screening information and education system will be implemented. The particularities of the index cases likely to require an adaptation of the device will be collected, analyzed and taken into account (level of health literacy, socio-economic status, level of education, professional activity ...). The analysis and intervention frameworks derived from theories on health behaviors will be mobilized (theory of reasoned action, theory of planned behaviors) and applied in order to reinforce the "intention" of the target audience. The analysis and intervention frameworks resulting from the educational sciences will be integrated with a "competence" approach (Aizen, 1991, Denovel, Dufour, Prochaska, 1983, Le Boterf, 2002).
  Arms: Therapeutic Education Strategy

SUMMARY:
The relative risk of colorectal cancer (CRC) is increased in first-degree relatives of patients with CRC or advanced adenoma. In the high-risk CCR population defined by a family history at the first stage of CRC or advanced adenoma before age 60, total colonoscopy is the recommended screening test. In France, the rate of screening colonoscopy in this population at high risk of CRC is insufficient, which limits the effectiveness of this targeted screening.

The main reason for this low participation rate is that most patients undergoing RCC or advanced adenoma are unaware of the family implications of their diagnosis and therefore reluctant to disseminate this information to their patients Related matters. The need for a better perception of the personal risk of CRC in first-degree relatives of patients with CRC or advanced adenoma, with the expected coronary adherence to increasing screening, requires a good understanding of risk through Clear, adapted and comprehensible information that can be relayed personally by the case-index.

The objective of this project is to develop a personalized prevention and screening program for the JRC in order to meet the needs of the relatives of the sick. The means of intervention that will be implemented respond to the need to better take into account the level of CRC risk in a family-based CRC screening and prevention approach adapted to a high-risk CRC group characterized by Family history at the first stage of CRC or advanced adenoma and, consequently, to improve the information of the subjects concerned by screening and prevention of CRC.

The aim of the case-index education is to induce its intervention with its relatives to promote CCR screening. The use of the index case, as a means of providing information to relatives, implies an educational and psychological approach, based on evidence, but adapted and personalized.

DETAILED DESCRIPTION:
The relative risk of colorectal cancer (CRC) is increased in first-degree relatives of patients with CRC or advanced adenoma. In the high-risk CCR population defined by a family history at the first stage of CRC or advanced adenoma before age 60, total colonoscopy is the recommended screening test. In France, the rate of screening colonoscopy in this population at high risk of CRC is insufficient, which limits the effectiveness of this targeted screening.

ELIGIBILITY:
List of inclusion criteria

Index case:

* Patients with colorectal adenocarcinoma or advanced adenoma diagnosed (definition of advanced adenoma (Winawer, 2006): adenoma of diameter ≥ 10 mm and / or severe dysplasia and / or with a villous contingent).
* Patients with at least one relative of the first degree belonging to the target population of the screening strategy evaluated (between 40 and 75 years of age and less than 10 years of age of the case-index) and residing in France.
* Affiliation of the patient to a social security scheme (including CMU).
* Understanding of the French language.

Related:

* They correspond to the target population at high risk of colorectal cancer targeted by this program of promotion of colonoscopy screening:
* Subjects related to 1st degree to the index case and in contact with it.
* Age between 40 and 75 years of age or less than 10 years of age of the index case.
* Resides in France

List of exclusion Criteria :

Index case :

* Chronic inflammatory bowel disease.
* Genetic predisposition syndrome identified with colorectal cancer (Lynch syndrome, familial polyposis linked to the APC and MYH genes).
* Patient's knowledge of a first-degree relative with colorectal adenocarcinoma or advanced adenoma.
* Isolated patient of his / her first-degree relatives and not wishing to re-establish contact with them.
* Advanced colorectal cancer with a life expectancy <6 months and / or a WHO ≥ 2 general condition.
* Transmission of information to the family already carried out.

Related :

- Not applicable

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
Participation rate in screening colonoscopy for first-degree relatives of patients with RCC or advanced adenoma. | 12 MONTHS
  Participation rate in screening colonoscopy for first-degree relatives of patients with RCC or advanced adenoma.

SECONDARY OUTCOMES:
Psychological determinants (quality of relationship with relatives, motivation to inform relatives) that can condition the enrollment in the education program. | 12 MONTHS
  Psychological determinants (quality of relationship with relatives, motivation to inform relatives) that can condition the enrollment in the education program.
Social and demographic factors in index cases associated with screening colonoscopy in related subjects: age, sex, educational level, socio-professional category. | 12 MONTHS
  Social and demographic factors in index cases associated with screening colonoscopy in related subjects: age, sex, educational level, socio-professional category.
Social and demographic factors associated with screening colonoscopy in related subjects: age, sex, educational level, socio-professional category. | 12 MONTHS
  Social and demographic factors associated with screening colonoscopy in related subjects: age, sex, educational level, socio-professional category.
How to access screening colonoscopy: pathway (public or private), direct access to the gastroenterologist or through the attending physician. | 12 MONTHS
  How to access screening colonoscopy: pathway (public or private), direct access to the gastroenterologist or through the attending physician.
Time to access the colonoscopy (time between the procedure and the completion of the screening colonoscopy). | 2 MONTHS
  Time to access the colonoscopy (time between the procedure and the completion of the screening colonoscopy).
Rate of colorectal cancer. | 12 MONTHS
  Rate of colorectal cancer.
Rate of advanced adenomas. | 12 MONTHS
  Rate of advanced adenomas.
Detection rate of scallop lesions. | 12 MONTHS
  Detection rate of scallop lesions.
Rate of complications in screening colonoscopies. | 12 MONTHS
  Rate of complications in screening colonoscopies.
Quality criteria for screening colonoscopy using the following parameters: visualization rate of the bottom of the colon, the withdrawal time of the colonoscope (Withdrawal time), quality of the colic preparation using the Boston scale. | 12 MONTHS
  Quality criteria for screening colonoscopy using the following parameters: visualization rate of the bottom of the colon, the withdrawal time of the colonoscope (Withdrawal time), quality of the colic preparation using the Boston scale.

CONTACTS AND LOCATIONS:
Overall Officials: CAROLI BOSC Françis- Xavier, Pr, Principal Investigator — University Hospital, Angers; MATYSIAK-BUDNIK Tamara, Pr, Principal Investigator — Nantes University Hospital; LANDAU Alain, Dr, Principal Investigator — CHG DREUX; GARGOT Denis, Dr, Principal Investigator — CHG BLOIS; BARBIEUX Jean- Pierre, Dr, Principal Investigator — CHG LOCHES; TOUGERON David, Pr, Principal Investigator — CHU Poitiers; LEGOUX Jean- Louis, Dr, Principal Investigator — CHR ORLEANS; BOURGEOIS Hugues, Dr, Principal Investigator — Clinic Victor Hugo LE MANS
Locations (8):
- France (8):
  - Service d'Hépatogastro-entérologie CHU ANGERS, Angers
  - Service d'Hépatogastro-entérologie CHG BLOIS, Blois
  - Service d'Hépatogastro-entérologie CHG de DREUX, Dreux
  - Service de Médecine CHG de Loches, Loches
  - Service d'Hépatogastro-entérologie CHU de NANTES, Nantes
  - Service d'Hépatogastro-entérologie CHR d'Orléans, Orléans
  - Service d'Hépatogastro-entérologie CHU POITIERS, Poitiers
  - Service d'Hépatogastro-entérologie CHRU de TOURS, Tours